CLINICAL TRIAL: NCT00468286
Title: An Open-Label, Multi-Centre, Randomised Parallel-Group Dose-Finding Study, Investigating Efficacy and Safety of Two Degarelix Three-Month Dosing Regimens in Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Brief Title: Investigating Efficacy and Safety of Two Degarelix Three-Month Dosing Regimens in Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS18
Record Dates: First submitted 2007-04-13; First posted 2007-05-02 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Treatment group A: Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 360 mg SC (by injection under the skin) given after 1, 4, 7, & 10 months.
  Interventions: Drug: Degarelix
- B (Experimental): Treatment group B: Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 480 mg SC (by injection under the skin) given after 1, 4, 7, & 10 months.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Experimental
  Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 360 mg SC (by injection under the skin) given after 1, 4, 7, & 10 months.
  Arms: A
Drug: Degarelix — Experimental
  Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 480 mg SC (by injection under the skin) given after 1, 4, 7, & 10 months.

SUMMARY:
The study will have two treatment groups, evaluating two Degarelix doses. First dose is the initial dose followed by a maintenance dose given every three months. The initial dose given to suppress the testosterone level and the three month maintenance dose to maintain the suppressed testosterone level over one year of treatment.

DETAILED DESCRIPTION:
An Open-Label, Multi-Centre, Randomized Parallel-Group Dose-Finding Study, Investigating Efficacy and Safety of Two Degarelix Three-Month Dosing Regimens in Patients with Prostrate Cancer Requiring Androgen Ablation Therapy.

ELIGIBILITY:
Inclusion / Exclusion Criteria:

* Patients, aged 18 years or older, with histologically proven prostate cancer of all stages in whom endocrine treatment is indicated.
* Screening testosterone level above the lower limit of normal range, globally defined as >2.2 ng/mL.
* Eastern Cooperative Oncology Group (ECOG) score of ≤2.
* Screening prostate-specific antigen (PSA) level ≥ ng/mL.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (29):
- United States (11):
  - Urology Centers of Alabama, Homewood, Alabama
  - South Orange County Medical Research Center, Laguna Woods, California
  - South Florida Medical Research, Aventura, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Regional Urology, Shreveport, Louisiana
  - Investigational site, Carmel, New York
  - The Urology Center, Greensboro, North Carolina
  - State College Urologic Association, State College, Pennsylvania
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Urology of Virginia Research, Norfolk, Virginia
  - Urology Research Center, Seattle, Washington
- Canada (4):
  - Investigational site, Surrey, British Columbia
  - Investigational site, Victoria, British Columbia
  - Investigational site, Kentville, Nova Scotia
  - The Female/Male Health Centres, Ontario
- Czechia (3):
  - Nemocnice Jindrichuv Hradec a.s., Hradec
  - Slezska nemocnice, Opava
  - Vseobecna fakultni nemocnice v Praze, Prague
- Hungary (4):
  - Dombóvári Szent Lukács Egészségügyi Kht, Dombóvár
  - Borsod-Abaúj-Zemplé n Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Miskolc Megyei Jogú Város Önkormányzat Miskolci Egészségügyi Központ, Miskolc
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Romania (7):
  - Private Medical Center, Arad
  - "Prof Dr Th Burghele" Clinical Hospital, Bucharest
  - Dinu Uromedica, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - E-Uro Medical Center S.R.L., Cluj-Napoca
  - Provita Center, Constanța
  - Sibiu County Clinical Hospital, Sibiu

RESULTS

PARTICIPANT FLOW:
Groups:
- Degarelix 240/360 mg: Treatment group A: Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 360 mg SC (by injection under the skin) given after 1, 4, 7, & 10 months.
- Degarelix 240/480 mg: Treatment group B: Initial dose of 240 mg SC (by injection under the skin) on day 0. Maintenance dose of 480 mg SC (by injection under the skin) given after 1, 4, 7, & 10 months.
Period: Overall Study
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Started | 67 (Started=Intention to treat (ITT) population.) | 66
Completed | 60 | 54
Not Completed | 7 | 12
Not completed — Adverse Event | 1 | 6
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg | Total
Number analyzed (Participants) | 67 | 66 | 133
Age Continuous [Mean (Standard Deviation); unit: years] — ITT population.
  years | 74.1 (7.3) | 72.7 (8.5) | 73.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT population.
  Participants
    Female | 0 | 0 | 0
    Male | 67 | 66 | 133
Race (NIH/OMB) [Count of Participants; unit: Participants] — ITT population.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 3 | 5
    White | 64 | 63 | 127
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram] — ITT population.
  kilogram | 78.9 (12.9) | 82.4 (13.4) | 80.6 (13.2)
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] — ITT population.
  kilogram per square meter | 27 (4.0) | 27.4 (3.4) | 27.2 (3.7)
Curative intent [Number; unit: participants] — ITT population. Curative intent refers to radical prostatectomy or radiotherapy.
  participants
    Yes | 7 | 6 | 13
    No | 60 | 60 | 120
Gleason Score [Number; unit: participants] — ITT population. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  Gleason score for 1 patient is missing
  participants
    2-4 | 8 | 3 | 11
    5-6 | 19 | 24 | 43
    7-10 | 39 | 39 | 78
    Data missing | 1 | 0 | 1
Stage of Prostate Cancer [Number; unit: participants] — ITT population. Stage of prostate cancer was classified according to the Tumour, Nodule and Metastatic classification that is a cancer staging system that describes the extent of cancer. T describes the size of the tumor and whether it has invaded nearby tissue, N describes regional lymph nodes that are involved, and M describes distant metastasis.
  participants
    Localized | 26 | 19 | 45
    Locally advanced | 17 | 22 | 39
    Metastatic | 14 | 16 | 30
    Not classifiable | 10 | 9 | 19
Time Since Prostate Cancer Diagnosis [Mean (Standard Deviation); unit: days] | 370 (1011) | 265 (499) | 319 (802)
Serum Testosterone [Median (Full Range); unit: ng/mL] — ITT population.
  ng/mL | 4.1 [2.0 to 10.4] | 4.1 [1.6 to 9.1] | 4.1 [1.6 to 10.4]
Serum PSA [Median (Full Range); unit: ng/mL] — ITT population.
  ng/mL | 22.9 [2.1 to 5309.6] | 18.2 [0.5 to 2668.4] | 20.3 [0.5 to 5309.6]
Serum FSH [Median (Full Range); unit: IU/L] | 8.4 [2.2 to 39.8] | 6.9 [1.6 to 52.2] | 7.0 [1.6 to 56.2]
Serum LH [Median (Full Range); unit: IU/L] | 5.9 [1.4 to 14.0] | 4.6 [1.9 to 34.0] | 5.3 [1.4 to 34.0]

OUTCOME MEASURES:

1. Primary Outcome: Probability of Testosterone at Castration Level (≤0.5 ng/mL) From Day 28 Through Day 364
Description: Kaplan-Maier estimates of the cumulative probabilities of testosterone <=0.5 ng/mL from Day 28 to Day 364.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
percentage of participants | 89.0 [78.3 to 94.6] | 93.3 [83.1 to 97.4]

2. Secondary Outcome: Serum Levels of Testosterone Over Time
Time Frame: 1 year
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
ng/mL
  Day 28 | 0.1 [0 to 0.5] | 0.1 [0 to 4.6]
  Day 84 | 0.1 [0 to 0.4] | 0.1 [0 to 1.1]
  Day 364 | 0.1 [0 to 2.4] | 0.1 [0 to 0.7]

3. Secondary Outcome: Probability of Testosterone at Castration Level (≤0.5 ng/mL) From Day 56 Through Day 364
Description: Kaplan-Maier estimates of the cumulative probabilities of testosterone <=0.5 ng/mL from Day 56 to Day 364.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
percentage of participants | 89.0 [78.3 to 94.6] | 93.3 [83.0 to 97.4]

4. Secondary Outcome: Probability of no PSA Failure
Description: Cumulative probability (%) and 95% confidence interval (CI) for completing the study without PSA failure. PSA failure was defined as two consecutive increases of 50%, and at least 5 ng/mL, compared to nadir (lowest level of PSA achieved).
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
percentage of participants | 93.5 [83.6 to 97.5] | 94.6 [84.3 to 98.2]

5. Secondary Outcome: Serum Levels of PSA Over Time
Time Frame: 1 year
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
ng/mL
  Day 28 | 3.5 [0 to 274.6] | 3.1 [0.2 to 91.3]
  Day 84 | 1.2 [0 to 37.2] | 1.2 [0 to 47.4]
  Day 364 | 0.4 [0 to 354.4] | 0.7 [0 to 135.5]

6. Secondary Outcome: Serum Levels of Follicle Stimulating Hormone (FSH) Over Time
Time Frame: 1 year
Measure: Median (Full Range); unit: IU/L
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
IU/L
  Day 28 | 0.3 [0.2 to 3.2] | 0.4 [0.2 to 8.1]
  Day 84 | 0.6 [0.2 to 3.9] | 0.5 [0.2 to 7.2]
  Day 364 | 1.6 [0.2 to 7.9] | 1.0 [0.2 to 9.2]

7. Secondary Outcome: Serum Levels of Luteinizing Hormone (LH) Over Time
Time Frame: 1 year
Measure: Median (Full Range); unit: IU/L
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
IU/L
  Day 28 | 0.1 [0 to 1.6] | 0.1 [0 to 4.7]
  Day 84 | 0.1 [0 to 1.4] | 0.1 [0 to 2.5]
  Day 364 | 0.3 [0 to 3.6] | 0.2 [0 to 2.1]

8. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal values in blood pressure (systolic and diastolic), pulse, and body weight during the trial. The table presents the number of participants with a normal baseline value and at least one post-baseline markedly abnormal value.
Time Frame: Baseline up to 1 year
Measure: Number; unit: participants
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 0
  Diastolic blood pressure >=105 and increase >=15 | 0 | 0
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 1 | 1
  Heart rate <=50 and decrease >=15 | 0 | 0
  Heart rate >=120 and increase >=15 | 0 | 0
  Body weight decrease of >=7 percent | 6 | 0
  Body weight increase of >=7 percent | 8 | 4

9. Secondary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Number analyzed (Participants) | 67 | 66
participants
  Abnormal alanine aminotransferase (ALAT) | 22 | 21
  Abnormal aspartate aminotransferase | 33 | 23
  Abnormal bilirubin | 3 | 1
  ALAT >3x upper limit of normal (ULN) | 1 | 3
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix 240/360 mg | Degarelix 240/480 mg
Serious Adverse Events (participants affected / at risk) | 7/67 | 11/66
Other Adverse Events (participants affected / at risk) | 49/67 | 53/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240/360 mg (N=67) | Degarelix 240/480 mg (N=66)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240/360 mg (N=67) | Degarelix 240/480 mg (N=66)
Injection site pain (General disorders) | 10 (19) | 13 (29)
Injection site erythema (General disorders) | 4 (4) | 5 (10)
Asthenia (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 5 (5)
Weight increased (Investigations) | 9 (9) | 5 (5)
Weight decreased (Investigations) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Testicular atrophy (Reproductive system and breast disorders) | 4 (4) | 4 (5)
Gynaecomastia (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Hot flush (Vascular disorders) | 24 (25) | 21 (23)
Hypertension (Vascular disorders) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.